CLINICAL TRIAL: NCT00979641
Title: Single Arm Study of the Combination of Biweekly Avastin and Docetaxel as the First Line Treatment for Patients With Metastatic Breast Cancer
Brief Title: Biweekly Avastin and Docetaxel as the First Line Treatment for Patients With Metastatic Breast Cancer
Acronym: AINO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Participants are no longer being examined. The results are published 2016 Anticancer Research 36: 6431-6438
Sponsor: Tampere University Hospital (Other)
Collaborators: Oulu University Hospital (Other); Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Pirkko-Liisa Kellokumpu-Lehtinen, professor of oncology and radiotherapy, Tampere University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2008-003527-24
Record Dates: First submitted 2008-12-19; First posted 2009-09-18 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Neoplasms
Keywords: breast cancer; metastatic; chemotherapy; bevacizumab; docetaxel; Phase II; first line chemotherapy; metastatic breast cancer patients
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Neoplasm Metastasis | interventions — Docetaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- chemoterapy (Experimental): docetaxel/paclitaxel + bevacizumab
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel
  Other Names: bevacizumab

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the combination of biweekly docetaxel and bevacizumab in the first line treatment of metastatic breast cancer by using Response Evaluation Criteria In Solid Tumors (RECIST criteria) and NCI Common Terminology Criteria for Adverse Events (NCI CTC-AE) version 3. In addition several biochemical makers are tested as possible predictive factors.

DETAILED DESCRIPTION:
Patients with histologically or cytologically proven measurable or nonmeasurable metastatic breast cancer are treated with a combination of biweekly docetaxel and bevacizumab as the first line treatment in multicenter phase II trial. The outcome measures would be PFS, Response rate (RECIST), duration of response, safety (NCI CTC-AE version 3) and survival. In addition several biochemical makers are tested as possible predictive factors. Treatment would be continued until PD, patient's refusal or treatment discontinuation due to side-effects or patients death. In responding patients bevacizumab would be continued either alone or in hormone receptor positive patients combined with hormone treatment until progression.

ELIGIBILITY:
Inclusion Criteria:

* written informed concent
* age > or equal 18 years
* able to comply with the protocol
* histologically or cytologically confirmed, Her-2 negative, adenocarcinoma of the breast with measurable or nonmeasurable metastatic disease, chemotherapy indicated
* ECOG 0-2, life expectancy of over or qual to 12 wks
* prior neo/adjuvant chemotherapy allowed
* prior adjuvant taxane therapy is allowed, DFS> or equal 6 months
* previous hormonal therapy allowed
* prior RT is allowed as adjuvant setting or to relief of metastatic bone pain, no more than 30% of marrow-bearing bone irradiated
* Adequate haematological function
* adequate liver function total bilirubin <1.5 x upper limit of normal and AST,ALT <2.5 x ULN in patients without liver metastases; <5 x ULN in patients with liver metastases
* adequate renal function serum creatinine <or equal 1,5x ULN or calculated creatinine clearance > or equal 50mL/min and urine dipstick for proteinuria <2+. Patients discovered to have or equal proteinuria or dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate < or equal 1 g of protein in 24 hours
* INR<or equal 1.5 and PTT< or equal 1.5 x ULN within 7 days prior to enrolment. Anticoagulation treatment not allowed
* if female, should not be pregnant or breast-feeding. Women with an intact uterus must have a negative serum pregnancy test within 28 days prior to inclusion into the study

Exclusion Criteria:

* previous chemotherapy for mBC
* radiation therapy for the treatment of metastatic disease within 28 days
* evidence of CNS metastases. If symptomatic, the patient should be scanned within 28 days to enrolment to rule out CNS metastases
* pre-existing peripheral neuropathy NCI CTC-AE grade > 2 at enrolment
* major surgery, significant traumatic injury within 28 days prior to enrolment or anticipation of the need for major surgery during study treatment
* Minor surgery, including insertion off an indwelling catheter, within 24 hours prior to the first line bevacizumab infusion
* Current or recent(within 10 daÿs of first dose of bevacizumab) use of aspirin (>325mg/day)
* current or recent (within 10 days of first dose of bevacizumab) use of oral or parenteral anticoagulants or thrombolytic agents.
* history of evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding
* uncontrolled hypertension (systolic >150mmHg and/or diastolic>100mmHg)
* Clinically significant cardiovascular disease for example CVA, myocardial infarction, unstable angina, congestive heart failure NYHA Class > or equal II, serious cardiac arrhythmia requiring medication during the study, which might interfere with regularity of the study treatment, or not controlled by medication
* non- healing wound, active peptic ulcer or bone fracture
* history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months of enrolment
* past of current history (within the last 5 years) of other malignancies except curatively treated basal and squamous cell carcinoma of the skin or in-situ carcinoma of the cervix
* treatment with any other investigational agent, or participation in another clinical drug trial within 28 days prior to enrolment
* evidence of any other disease, neurological, psychiatric or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications
* history of thrombotic disorders within last six months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
progression free survival | 1-3 months
  increase of cancer burden

SECONDARY OUTCOMES:
efficacy, changes in metastacic lesions | every 2 months
  response rate
overall survival | 2- 3 months
  alive
time to response | 2 months
  decrease of cancer burden
duration of response | 2 months
  gain
progression free survival from first relapse | 2 months
  second increase of cancer burden
safety, occurence of side-effects | 1 month
  side effects according to NCICTC-AE version 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Pirkko-Liisa I Kellokumpu-Lehtinen, MD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere Unviersity Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maenpaa N, Tiainen L, Hamalainen M, Luukkaala T, Tanner M, Lahdenpera O, Vihinen P, Karihtala P, Kellokumpu-Lehtinen PL, Moilanen E, Jukkola A. Neuropilin-1 and placental growth factor as prognostic factors in metastatic breast cancer. BMC Cancer. 2024 Mar 11;24(1):331. doi: 10.1186/s12885-024-12070-7. PMID 38468231
- [Derived] Tiainen L, Korhonen EA, Leppanen VM, Luukkaala T, Hamalainen M, Tanner M, Lahdenpera O, Vihinen P, Jukkola A, Karihtala P, Aho S, Moilanen E, Alitalo K, Kellokumpu-Lehtinen PL. High baseline Tie1 level predicts poor survival in metastatic breast cancer. BMC Cancer. 2019 Jul 24;19(1):732. doi: 10.1186/s12885-019-5959-8. PMID 31340773
- [Derived] Tiainen L, Tanner M, Lahdenpera O, Vihinen P, Jukkola A, Karihtala P, Paunu N, Huttunen T, Kellokumpu-Lehtinen PL. Bevacizumab Combined with Docetaxel or Paclitaxel as First-line Treatment of HER2-negative Metastatic Breast Cancer. Anticancer Res. 2016 Dec;36(12):6431-6438. doi: 10.21873/anticanres.11241. PMID 27919965
- Available data/document: Clinical Study Report — http://www.anticancerresearch.com